CLINICAL TRIAL: NCT06410625
Title: Evaluation of the Response to Chemo-Therapy by FLT PET in Mesothelioma
Brief Title: Evaluation of Response by FLT PET in Mesothelioma
Acronym: FLT-MM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Collaborators: Liv Hospital Ankara (Other); Ankara Yildirim Beyazıt University (Other); Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Cigdem Soydal, Asc Prof of Nuclear Medicine, Ankara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLT-MM
Record Dates: First submitted 2024-03-27; First posted 2024-05-13 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Pleural Mesothelioma; Treatment Response; Chemotherapy Effect
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Patients who will receive standardized chemotherapy for pleural mesothelioma
  Interventions: Diagnostic Test: FLT PET imaging

INTERVENTIONS:
Diagnostic Test: FLT PET imaging — Evaluation of response to chemotherapy with FLT PET imaging
  Other Names: FDG PET

SUMMARY:
Pleural mesothelioma (MPM) is an aggressive tumor that affects the pleura and originates from mesothelial cells. If untreated, median survival is 4-12 months following diagnosis. Asbestos exposure is a risk factor associated with 80% of cases. After the 1980s, regulations controlling the use of asbestos ensured that cases were limited. Approximately 3,000 new cases are diagnosed each year in the United States. In general, a minority of patients are candidates for surgery at the time of presentation, so the mainstay of treatment is systemic chemotherapy. For patients who are surgical candidates, surgery is usually part of a multimodal treatment process that also includes chemotherapy and/or radiotherapy. Early and accurate diagnosis has a critical impact on the management of the disease due to limited response to multimodal treatments. Patients are often diagnosed at an advanced stage, leading to poor overall survival. Thorax and upper abdomen CT imaging are standard initial imaging modalities for clinical staging of MPM. Although CT identifies the general extent of the primary tumor, it may not definitively identify some areas of tumor invasion. There may be difficulties especially in the evaluation of chest wall and diaphragm invasion.

18F-FDG PET/CT has been widely used for cancer diagnosis, staging, treatment response and prognostic information for many years with high accuracy rates. 18F-FDG PET/CT provides valuable information on differentiating benign and malignant pleural abnormalities, evaluating the possibility of malignant involvement of mediastinal and hilar lymph nodes, and detecting distant metastases. 18F-FDG PET/CT identifies metastatic disease undetected on CT in approximately 10% of patients. At the same time, the degree of involvement (SUV) in FDG PET plays a role in predicting disease prognosis. 18F-FDG PET/CT can also be used to evaluate the treatment response in patients receiving chemotherapy, but due to chemotherapy-related inflammatory changes, it is necessary to wait at least 2 weeks to evaluate the treatment response.

18F-Fluorothymidine (FLT) is a thymidine kinase 1-specific substrate that is increased in proliferating cells and is associated with the Ki-67 index, a proliferation marker. It allows noninvasive evaluation of cell proliferation, especially the early evaluation of the response to cytotoxic chemotherapy. 18F-FLT PET/CT imaging has shown success in early evaluation of response to systemic endocrine, chemotherapy, radiotherapy and combined chemotherapy in multiple tumor types. The prognostic value of a decrease in 18F-FLT uptake after initiation of treatment has also been reported.

In this study, it is aimed to evaluate the success of 18F-FLT PET/CT in the early evaluation of the response after the first cycle of chemotherapy in patients diagnosed with mesothelioma and receiving systemic chemotherapy. It is also aimed to evaluate the prognostic value of response evaluation made with this method.

It is planned to prospectively include 25 patients with MPM who scheduled for chemotherapy in the study. Included patients will undergo 18F-FDG PET/CT before chemotherapy followed by 18F-FLT PET/CT imaging within two weeks. 18F-FLT PET/CT will be performed on the 4th day after the 1st cycle of chemotherapy. After chemotherapy is completed, treatment response will be evaluated with 18F-FDG PET/CT. Patients will then be followed by their clinicians for relapse and progressive disease. Thus, the success of early 18F-FLT PET/CT in predicting end of treatment response will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Having a histopathologically confirmed diagnosis of Pleural Mesolthelioma
* Patients planned for platinum-based chemotherapy
* Patients who gave informed consent form to participate in the study

Exclusion Criteria:

* Being under 18 years old
* Patients planned for immunotherapy
* Patients who did not provide informed consent form to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
The early treatment response by FLT PET | 1-4 days
  Evaluation of the response to chemotherapy with change in the uptake of FLT in PET in pleural mesothelioma patients

SECONDARY OUTCOMES:
The prognostic importance of treatment response evaluated with FLT PET | 1 year
  Evaluation of the predictive value for progression free survival and overall survival of FLT PET reponse after chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Medical School, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No